CLINICAL TRIAL: NCT05194527
Title: The Detrimental Course of Acute Intestinal Ischemia: Improvement of the Diagnosis
Brief Title: The Detrimental Course of Acute Intestinal Ischemia
Acronym: TACTIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University (Other)
Collaborators: Maastricht University Medical Center (Other); Gelre Hospitals (Other); Medisch Spectrum Twente (Other); University Medical Center Groningen (Other); Universitaire Ziekenhuizen KU Leuven (Other); Amsterdam UMC (Other); Maag Lever Darm Stichting (Other)
Responsible Party: Sponsor
Other Study IDs: TACTIC study
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Diagnoses Disease; Acute Mesenteric Ischemia; Intestinal Disease
Keywords: Acute Mesenteric Ischemia; Volatile Organoic Compounds; Plasma/Serum Biomarkers; SM22; Villin-1; I-FABP; Diagnosis
MeSH Terms: conditions — Intestinal Diseases; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — After patient inclusion, blood and air samples will be collected at consecutive time points. Plasma will be isolated from the collected blood and analyzed by enzyme-linked immunosorbent assay (ELISA) for the selected biomarkers: I-FABP, SM22 and VIL-1. ELISAs for I-FABP, Exhaled air will be stabilized on carbon desorption tubes until analysis. The VOC profile will be analyzed by gas chromatography time of flight mass spectrometry (GC-TOF-MS) including compound separation by GC and full mass spectra recording by TOF-MS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Acute Mesenteric Ischemia: Patients that are diagnosed with Acute mesenteric Ischemia
  Interventions: Other: Biomarker validation and VOC profile identification
- Patient with another underlying disease/condition: Patients that are diagnosed not with acute mesenteric ischemia, but with a other underlying disease/condition
  Interventions: Other: Biomarker validation and VOC profile identification

INTERVENTIONS:
Other: Biomarker validation and VOC profile identification — Validation of a panel of plasma markers for the early diagnosis of acute intestinal ischemia with a panel consists of I-FABP, VIL-1, and SM22. Identification of an acute intestinal ischemia specific VOCs profile and evaluate exhaled breath analysis as a diagnostic tool for intestinal ischemia.

SUMMARY:
Rationale:

Acute intestinal ischemia is a life-threatening condition with a short-term mortality that can range up to 80%. Medical diagnosis and treatment have remained troublesome, due to the clinical presentation which is mostly characterized by non-specific signs and symptoms. Early unambiguous diagnosis of acute intestinal ischemia is critical to prevent progression from reversible to irreversible intestinal injury, and henceforth decrease morbidity and improve survival.

Objective:

We aim to validate a panel of plasma biomarkers and investigate volatile biomarkers that allow early and accurate identification of acute intestinal ischemia in patients. In addition, we aim to identify a volatile organic compound (VOC) profile specific for acute intestinal ischemia in exhaled breath.

Study design: Prospective observational study

Study population:

All patients suspected of acute intestinal ischemia Main study parameters: The primary endpoint of the study is the early and accurate identification of presence and severity of acute intestinal ischemia in patients. The main study parameters are plasma biomarkers indicative for intestinal damage and volatile organic compounds (VOC) in exhaled air of patients suspected of acute intestinal ischemia.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

There is a minimal amount of risks involved in participating in this study. Blood samples will be obtained with the use of an arterial line, intravenous line (IV), central venous catheter (CVC), peripheral venous catheter (PVC) or a venepuncture. The risk of venepuncture is a small local hematoma. In addition to blood sampling, we will also obtain exhaled air. This non-invasive procedure takes approximately 5 minutes in which patients breath in a 3L Tedlar bag at a normal frequency and volume. This procedure will not cause any physical strain. Collection of samples and data will take place during the hospital stay of the included patients. For this reason, no additional hospital visits are required for this study. Participating patients in this study will have no direct benefits, but in the future the results of our study will likely be useful in the early diagnosis of patients suspected of acute intestinal ischemia.

The research goal in this study is the early identification of patients that suffer from acute intestinal ischemia. These patients are difficult to diagnose due to a multitude of non-specific symptoms and the lack of fast and specific tests. In this study we will be able to investigate patients that are admitted with acute abdominal complications and observe them in the early stages of their condition. Accordingly, we will be able to evaluate the proposed panel of biomarkers and to identify VOC patterns in patients with acute abdominal complications.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE Acute intestinal ischemia remains a common clinical emergency with short-term mortality up to 80% and is often highly underestimated. , , It is a life-threatening clinical condition of diminished blood flow towards the gut, resulting in decreased supply of oxygen and nutrients to the intestinal tissue. Prolonged periods of ischemia are associated with disruption of the intestinal wall that normally functions as an important barrier. , The intestinal wall is composed of different layers and has a multitude of functions, such as the absorption of nutrients as well as the protection against harmful pathogens and carcinogens located in the intestinal lumen. When tissue damage occurs as consequence of ischemia, it progresses from the inner to the outer intestinal layer. This event results in release of a specific set of structural and functional proteins. Over the past few years many circulating biomarkers, such as D-dimer, glutathione S-transferase (GST), D-lactate and citrulline have been described as potential biomarkers for intestinal ischemia , , .

The incidence of acute intestinal ischemia increases exponentially with age, with an equal occurrence between men and women. Consequently, it is expected that there will be a strong increase in the incidence of acute intestinal ischemia due to population aging. Once there is a high index of suspicion of acute intestinal ischemia, the clinician should act fast. Early unambiguous diagnosis of the ischemic intestine is crucial to prevent further progression from reversible to irreversible intestinal injury, and henceforth decrease morbidity and mortality.

Despite the advances in medical diagnosis and treatment over the past decades, intestinal ischemia still has a poor prognosis.1 Delayed diagnosis is one of the leading causes of the high mortality rates. Delayed recognition of this condition results into the development of irreversible intestinal necrosis- and peritonitis, which is closely correlated with the high mortality in these patients. There are various causes of intestinal ischemia, which are generally divided into two categories: causes of vascular origin (mesenteric embolism/thrombosis, or non-occlusive mesenteric ischemia) and non-vascular causes (such as strangulated intestinal obstruction). Interestingly, there is a high variation of clinical presentation and features between the various causes of acute intestinal ischemia. The clinical presentation is mostly characterized by non-specific signs and symptoms for instance, abdominal pains, loss of weight, elevated blood cell count and metabolic acidosis.1-3, For example, arterial embolisms are associated with nausea and vomiting, whereas, thrombotic mesenteric arterial occlusion is more commonly associated with pain that intensifies after food ingestion .

Currently, high-tech diagnostic equipment such as compute tomography (CT) imaging is used for diagnosis. However, identification of acute intestinal ischemia by CT remains difficult, because most of the characteristic features such as occlusion of mesenteric vessels, bowel wall thickening and intestinal pneumatosis can be easily missed. , , Also, these features are highly variable and non-specific, i.e. they overlap with radiological appearances of other acute abdominal complications. It remains a challenge, even for experienced clinicians, to identify patients who are at risk of acute intestinal ischemia among patients presenting with other conditions. Hence, fast and accurate diagnosis is vital for improving the clinical outcomes of patients with acute intestinal ischemia.

In recent years, a number of studies have described new potential biomarkers, such as intestinal fatty acid binding protein (I-FABP), for the identification of acute intestinal ischemia. Previously, it has been shown in our lab that I-FABP plasma levels are increased in patients suffering from intestinal ischemia. I-FABP is a small (14-15 kDa) intracellular and water-soluble protein that is specifically expressed by mature epithelial cells in the intestinal mucosa. I-FABP has a high abundancy within the small intestine and accounts for approximately 2% of the cytosolic protein expressed. , Upon a decrease of bowel perfusion and consequent loss of enterocyte cell membrane integrity, a rapid release of I-FABP within the circulation is observed. In an earlier study, we could reveal a relationship between the release of I-FABP and the severity of intestinal ischemia mucosal damage, where I-FABP levels in the circulation were inversely correlated with the remaining villus length. The exclusive expression of I-FABP in the intestine potentially makes it an important marker for the early detection of intestinal damage as a consequence of ischemia.

Another biomarker of intestinal ischemia is the cytoskeleton protein Villin-1 (VIL-1). VIL-1 is a large (95 kDa) protein that is localized in the cytoplasm and luminal membranes where it is described to play a role in actin regulation. , It was shown in rat and human models of ischemia that VIL-1 is released into the circulation and can be measured in plasma (Ceulemans et al. submitted, 2018). As opposed to I-FABP, VIL-1 remained detectable during prolonged periods after the onset of ischemic damage in rats due to the longer half-life. Plasma protein levels of VIL-1 correlated strongly with histopathological damage scored according to Park-Chiu. , I-FABP disappears after 30 minutes of reperfusion, whereas serological VIL-1 levels persist relatively high until 120 minutes after onset of reperfusion. Thus, these data indicate that both I-FABP and VIL-1 may provide new information on the duration of the ischemic events in humans.

Ischemia can cause significant damage to the mucosal layer within a short amount of time. Fifteen minutes of ischemia results into the formation of sub-epithelial spaces (a.k.a. 'blebs'), whereas ischemic periods lasting longer than 45 minutes can lead to irreversible mucosal damage.23, , Sustained periods of ischemia result in damage to the muscle layers also known as transmural ischemia. Transmural ischemia can develop into perforation of the intestinal wall, sepsis and eventually death.2, Plasma I-FABP and VIL-1 are very sensitive biomarkers for the identification of early intestinal mucosal damage. Adding a smooth muscle marker, such as Smooth Muscle 22 (SM22) to the panel of biomarkers could aid in evaluating the severity of the transmural ischemic tissue damage. SM22 is a small (22 kDa), water-soluble protein that is abundantly expressed in intestinal smooth muscle cells. , An experimental rat model revealed that SM22 is rapidly released in plasma upon ischemic damage, and remains detectable up to 6 hours following the induction of ischemia. Histology revealed complete disintegration of the villi following 4 hours of ischemia. Furthermore, immunohistochemical staining for SM22 indicated necrosis of the longitudinal muscle layer of the intestinal wall after 4 hours of ischemia, demonstrating that there is a transition from mucosal damage into transmural damage in this period of time. In patients with proven transmural infarction, SM22 plasma levels were significantly higher compared to patients with only mucosal ischemic injury or healthy controls.33 In addition, it was demonstrated that SM22 plasma levels were significantly higher in patients suffering from ischemia compared with patients that had other acute abdominal complaints. These data indicate that SM22 is most certainly a relevant biomarker to evaluate the severity of acute intestinal ischemia.

The last part of this study focuses on the analysis of volatile organic compounds (VOCs) in exhaled air of patients suspected of acute intestinal ischemia. The many hundreds of VOCs in exhaled air can give valuable information about several processes, such as metabolism and lipid peroxidation. The analysis of VOCs in exhaled air is a non-invasive technique that can be used to differentiate between various clinical conditions. Our project group already demonstrated the capability of VOC profiling to discriminate patients with intestinal and liver diseases such as inflammatory bowel disease (IBD) and non-alcoholic steatohepatitis from healthy subjects. , , Furthermore, chemical identification of VOCs from patients with Crohn's disease revealed that VOCs are involved in inflammatory, oxidative stress, gut barrier and leaky gut processes (Smolinska A, et al. in preparation). As the pathophysiologic processes of IBD and intestinal ischemia share common mechanisms, it is expected that VOC analysis will aid in the diagnosis of intestinal ischemia in a non-invasive manner. In a pilot study, we demonstrated that systemic inflammatory responses triggered by circulating endotoxin in human volunteers could be accurately detected using VOCs (Figure 2, Lubbers et al. in preparation). As VOC analyses can detect changes in metabolic and inflammatory processes with a high sensitivity and specificity, this promising technique enables early detection of the pathophysiologic processes occurring in intestinal ischemia. Altogether, these findings support the hypothesis that VOC profiles improve the diagnosis of intestinal ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* All consecutive patients admitted to one of the participating medical centers emergency departments (ED) or at the intensive care unit (ICU) (see 4.1 Population Base) with clinical suspicion of acute intestinal ischemia, which is based on;

  * clinical manifestation;
  * physical examination by the physician;
  * laboratory measurements;
  * physician's consideration to perform computed tomography (CT)-scan

Exclusion Criteria:

A subject who meets any of the following criteria will be excluded from participation in this study:

* Age ≤ 18 years In order to evaluate the performance of the panel of markers for the acute intestinal ischemia in clinical practice, the study population must resemble the clinical patient population as closely as possible

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients, clinically suspected of intestinal ischemia attending Maastricht University Medical Centre+ (MUMC+, Maastricht, The Netherlands), Amsterdam UMC (VUmc/AMC, Amsterdam, The Netherlands), Gelre Ziekenhuizen Apeldoorn (Apeldoorn, The Netherlands), Medisch Spectrum Twente (MST, Enschede, The Netherlands), University Medical Centrum Groningen (UMCG) and University Hospitals Leuven (UZ, Leuven, Belgium). The clinical course of all patients will be monitored. Diagnosis of intestinal ischemia will be based on findings from physical examination, laboratory measurements, surgery or autopsy, and verified by histopathological examination of the intestine by experienced pathologists, as well as evaluation of computed tomography (CT) scans.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
The main study parameters are plasma biomarkers indicative for intestinal damage of patients suspected of acute intestinal ischemia. | Inclusion (T0 min), 60 min (T60), 120 min (T120), 180 min (T180), Preoperative (PREOP), Reperfusion (RPF), Day 1 (T1), Day 2 (T2), Day 3 (T3), Day 4 (D4), Day 5 (D5)
  The primary outcome parameter in this study is the optimal cut-off values (from the combined plasma biomarkers) for classifying clinical cases that are positive or negative for acute intestinal ischemia.

SECONDARY OUTCOMES:
Secondary parameters in this study are the expression of VOCs in exhaled air of patients suspected of acute intestinal ischemia. | Inclusion (T0 min), 60 min (T60), 120 min (T120), 180 min (T180), Preoperative (PREOP), Reperfusion (RPF), Day 1 (T1), Day 2 (T2), Day 3 (T3), Day 4 (D4), Day 5 (D5)
  The secondary outcome in this study is the identification of specific VOC profiles for ischemia vs. non-ischemia patients. The individual compounds of this VOC profile are identified in order to discover novel pathophysiologic pathways involved in intestinal ischemia

CONTACTS AND LOCATIONS:
Overall Officials: Annet Duivenvoorden, MSc, Study Chair — Maastricht University; Kaatje Lenaerts, PhD, Principal Investigator — Maastricht University
Locations (6):
- Universitair Ziekenhuis Leuven, Leuven, Vlaams-Brabant, Belgium
- Netherlands (5):
  - Gelre Ziekenhuizen, Apeldoorn, Gelderland
  - Maastricht University Medical Centre+ (MUMC=), Maastricht, Limburg
  - Amsterdam University Medical Centre (UMC) - Location VUMC, Amsterdam, North Holland
  - Amsterdam University Medical Centre (UMC) - Location AMC, Amsterdam, North Holland
  - University Medical Centre Groningen (UMCG), Groningen

IPD SHARING:
Plan to Share IPD: Undecided
Uncertain

REFERENCES:
- [Derived] Duivenvoorden AAM, Clarysse M, Ceulemans LJ, Geelkerken RH, Derikx JPM, de Vries JPM, Buscher HCJL, Olde Damink SWM, van Schooten FJ, Lubbers T, Lenaerts K; Dutch Mesenteric Ischemia Study group (DMIS). Diagnostic potential of plasma biomarkers and exhaled volatile organic compounds in predicting the different stages of acute mesenteric ischaemia: protocol for a multicentre prospective observational study (TACTIC study). BMJ Open. 2023 Aug 29;13(8):e072875. doi: 10.1136/bmjopen-2023-072875. PMID 37643848
- See also: Continuous administration of enteral lipid- and protein-rich nutrition limits inflammation in a human endotoxemia model — https://pubmed.ncbi.nlm.nih.gov/23388517/
- See also: Early diagnosis of intestinal ischemia using urinary and plasma fatty acid binding proteins — https://pubmed.ncbi.nlm.nih.gov/21245670/
- See also: Plasma intestinal fatty acid-binding protein levels correlate with morphologic epithelial intestinal damage in a human translational ischemia-reperfusion model — https://pubmed.ncbi.nlm.nih.gov/24100750/
- See also: Human intestinal ischemia-reperfusion-induced inflammation characterized: experiences from a new translational model — https://pubmed.ncbi.nlm.nih.gov/20348235/
- See also: SM22 a Plasma Biomarker for Human Transmural Intestinal Ischemia — https://pubmed.ncbi.nlm.nih.gov/28525410/
- See also: Acute mesenteric ischemia: a clinical review — https://pubmed.ncbi.nlm.nih.gov/15159262/